CLINICAL TRIAL: NCT06765850
Title: Measurement of the Metabolome in Melanoma Patients Using NMR Spectroscopy and Gas Chromatography.
Brief Title: The Study Aims to Measure the Metabolome in Melanoma Patients Using NMR Spectroscopy and Gas Chromatography and to Analyse Differences Depending on the Course of the Disease.
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: University Hospital Carl Gustav Carus (Other)
Responsible Party: Principal Investigator, Frank Friedrich Gellrich, Senior Physician in Dermatology and Medical Tumor Therapy, Principal Investigator, MD, University Hospital Carl Gustav Carus
Other Study IDs: Melanomix
Record Dates: First submitted 2024-12-17; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Melanoma of Skin
Keywords: Melanoma; Metabolomics; NMR
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, various body fluids and tumour tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective, single-centre study with the central question of how the metabolome from blood samples, different body fluids and tissues between patients patients with malignant melanoma in different tumour tumour stages and healthy patients and whether this is suitable for early detection of initial diagnosis, recurrence or stage shift at an early stage.

The biosamples are collected in the BioBank Dresden and used for the NMR and LC-MS analyses described here. It is planned to use the biosamples for further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Current or past history of melanoma
* Ongoing therapy or tumour aftercare at the Skin Cancer Centre at Dresden University Hospital

Exclusion Criteria:

* Refusal to participate in the study
* Lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving ongoing tumour therapy or tumour aftercare at the Skin Cancer Centre at Dresden University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Differences in metabolite concentrations | through study completion, an average of 3 years
  Metabolite concentrations are measured by NMR spectroscopy and gas chromatography and compared between different subgroups.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Carl Gustav Carus, Dresden, Saxony, Germany